CLINICAL TRIAL: NCT03396523
Title: Losartan Effects on the Extinction of Conditioned Fear in Humans
Brief Title: Losartan and Emotion Processing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Benjamin Becker, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-25
Record Dates: First submitted 2018-01-04; First posted 2018-01-11 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Healthy
Keywords: Losartan; Fear extinction
MeSH Terms: interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Losartan group (Experimental)
  Interventions: Drug: Losartan
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Losartan — administration of losartan (50 mg) (oral)
  Other Names: Cozaar Oral Tablet
  Arms: Losartan group
Drug: Placebo Oral Tablet — administration of placebo (oral)
  Arms: Placebo group

SUMMARY:
The aim of the study is to investigate the effect of losartan (50mg, single dose) on the extinction of conditioned fear

DETAILED DESCRIPTION:
In a double-blind, between-subject, placebo controlled design the effects of a single dose of losartan (50mg) on fear extinction in healthy male participants will be examined. Participants will initially undergo a Pavlovian fear conditioning procedure, followed by the administration of 50mg losartan or placebo. 90 minutes after treatment subjects will undergo the fear extinction procedure. Neural activity and psychophysiological indices of arousal will be assessed by the simultaneous acquisition of functional magnetic resonance imaging (fMRI) and skin conductance data.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without past or current psychiatric or neurological disorders

Exclusion Criteria:

* history of head injury
* medical or psychiatric illness
* hypertension

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-01-04 (Actual); Primary Completion 2018-10-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Losartan effects on neural activity during fear extinction | 1 hour
  Neural activity will be measured by functional magnetic resonance imaging (fMRI). Effects of treatment will be evaluated by comparing extinction-related neural activity in the core extinction network (prefrontal cortex, limbic regions) between the active treatment and the placebo group.

SECONDARY OUTCOMES:
Losartan effects on skin conductance responses during fear extinction | 1 hour
  Effects of treatment will be evaluated by comparing extinction-related skin conductance responses between the active treatment and the placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Becker, PhD, Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- University of Electronic Science and Technology of China, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou F, Geng Y, Xin F, Li J, Feng P, Liu C, Zhao W, Feng T, Guastella AJ, Ebstein RP, Kendrick KM, Becker B. Human Extinction Learning Is Accelerated by an Angiotensin Antagonist via Ventromedial Prefrontal Cortex and Its Connections With Basolateral Amygdala. Biol Psychiatry. 2019 Dec 15;86(12):910-920. doi: 10.1016/j.biopsych.2019.07.007. Epub 2019 Jul 25. PMID 31471037